CLINICAL TRIAL: NCT00807716
Title: The Immediate and Long Term Effects of a Walking-skill Program Compared to Usual Physiotherapy Care in Patients Who Have Undergone Total Knee Arthroplasty (TKA): A Randomized Controlled Trial
Brief Title: Effect of Physiotherapy After Total Knee Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oslo (Other)
Responsible Party: Principal Investigator, Vigdis Bruun-Olsen, PHD student, University of Oslo
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2008/2436
Record Dates: First submitted 2008-12-11; First posted 2008-12-12 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-12

CONDITIONS: Knee Osteoarthritis
Keywords: physiotherapy; functional outcome; activity level; self efficacy; task oriented exercises
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- walking skill group (Experimental): weight-bearing 12 times, 70 minutes
  Interventions: Other: walking skill group
- usual physiotherapy care (Active Comparator): partial weight-bearing, 12 times, 40 minutes
  Interventions: Other: usual physiotherapy care

INTERVENTIONS:
Other: walking skill group — 12 Individualized group training sessions with focus on functional exercises like walking and stair climbing including balance training under physiotherapy guidance, 12 times 70 minutes.
  Arms: walking skill group
Other: usual physiotherapy care — physiotherapy, mostly in non-weight bearing, 12 times 40 minutes
  Arms: usual physiotherapy care

SUMMARY:
Physiotherapy plays an important part in rehabilitation after total knee arthroplasty. Even if this is a common practice, few studies have been performed on this issue.

The prime aim of this study is to examine the effects of an ambulatory individualized task-oriented exercise program compared with current ambulatory physiotherapy(usual care)on activity performance and self efficacy beliefs in the time span 6 weeks to 3 months after total knee arthroplasty with a follow-up at twelve months.

HO:Task oriented physiotherapy has better effect than usual care on activity performance and self-efficacy beliefs in the time span 6 weeks to 3 months after total knee replacement.

DETAILED DESCRIPTION:
A randomized controlled trial was performed with an experiment group having task oriented exercises in only weight-bearing 12 times from 6 weeks to 12 weeks after the operation, while the control group had usual physiotherapy care during the same time span. The primary outcome was walking measured by the six minutes walk test. Other performed and self reported measures of physical functioning were performed, at baseline, six weeks after the operation, immediately after the intervention at 12-14 weeks and with a follow-up nine months after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Primary gonarthrosis
* Good written and oral understanding of Norwegian
* Good cognitive function

Exclusion Criteria:

* Severe gonarthrosis in the other knee or coxarthrosis
* Neurological disorders or rheumatoid arthritis

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2008-10; Primary Completion 2010-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
6 minutes walk test | preoperatively, baseline at 6 weeks, after the intervention at 3 months, 12onths

SECONDARY OUTCOMES:
Self reported pain and activity level(KOOS) | preoperatively, 6 weeks, 3 months and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Anne Marit Mengshoel, PhD, Study Director — professor
Locations (1):
- Section of Nursing and Health Science, University of Oslo, Oslo, Norway